CLINICAL TRIAL: NCT03562507
Title: ERICA: Phase 2 Multi-center Trial of ESK981 in Combination With Nivolumab in Patients With Metastatic Renal Cell Carcinoma
Brief Title: Multi-center Trial of ESK981 in Combination With Nivolumab in Patients With Metastatic Renal Cell Carcinoma
Acronym: ERICA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of patient population
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2018.052; HUM00142975 (Other: University of Michigan)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Results first posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Renal Cell Carcinoma, Metastatic
Keywords: ESK981
MeSH Terms: conditions — Carcinoma, Renal Cell; Neoplasm Metastasis | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: There are 2 cohorts for accrual with Cohort A being accrued first. Cohort B will follow and will have 2 stages of accrual. Cohort A will accrue 11 patients to monotherapy treatment. Then Cohort B will begin accrual of 17 patients to the first stage and if the interim permits, the second stage will accrue an additional 19 patients.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ESK981 Monotherapy (Experimental): ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Interventions: Drug: ESK981
- ESK981 and Nivolumab (Experimental): ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Nivolumab: 480 mg/dose IV, Day 1 of each 28-day cycle
  Interventions: Drug: ESK981; Drug: Nivolumab

INTERVENTIONS:
Drug: ESK981 — ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
Drug: Nivolumab — 480 mg/dose IV, Day 1 of each 28-day cycle
  Arms: ESK981 and Nivolumab

SUMMARY:
The objective of the trial is to determine the clinical efficacy of ESK981 in combination with nivolumab therapy in patients with metastatic renal cell carcinoma (RCC).

DETAILED DESCRIPTION:
The study was terminated early due to changes in the RCC treatment landscape which limited the patient population. Due to this early termination no subjects were enrolled into Cohort B.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of renal cell carcinoma (any histology except medullary carcinoma or collecting duct carcinoma is acceptable) with radiologic or histologic evidence of metastatic disease.
* Prior treatment with up to one (and only one) anti-VEGF or VEGFR inhibitor (small molecule or antibody).
* Must have measurable disease as per Response Evaluation Criteria in Solid Tumors, version 1.1 (RECIST 1.1) criteria.
* Must be of age ≥ 18 years at time of informed consent.
* Ability to understand and the willingness to sign a written informed consent.
* Karnofsky Performance Status ≥60. (The Karnofsky Performance Status Scale is an assessment tool for functional impairment. It can be used to compare effectiveness of different therapies and to assess the prognosis in individual patients. In most serious illnesses, the lower the Karnofsky score, the worse the likelihood of survival.)
* Most recent systemic therapy or most recent radiation therapy ≥ 2 weeks of first study drug dose.
* Recovery to baseline or < Grade 1 CTCAE v.4.03 from toxicities related to any prior treatments, unless AE(s) are clinically non-significant and/or stable on supportive therapy.
* Women of childbearing potential must have a negative serum or urine pregnancy test within 28 days prior to registration.
* Adequate organ and marrow function

Exclusion Criteria:

* Prior treatment for metastatic disease with >1 anti-VEGF/VEGFR inhibitor.
* Prior treatment with anti-PD/PD-L1/CTLA4/IDO antibody (for Cohort B patients only) or ESK981 (for Cohort A and Cohort B patients).
* Prior mTOR inhibitors or glutaminase inhibitors are allowed.
* Untreated brain metastases or spinal cord compression.
* Uncontrolled hypertension defined as blood pressure >150/90 despite at least 2 anti-hypertensive medication(s) as assessed by 2 blood pressure readings taken at least 1 hour apart during screening.
* Major surgical procedure or significant traumatic injury within 6 weeks prior to study registration (> 6 weeks prior to registration is permitted as long as they have fully recovered from any such procedure).
* History of another primary malignancy except for: malignancy treated with curative intent and no known active disease for ≥2 years, adequately treated non-melanoma skin cancer without current evidence of active disease, adequately treated carcinoma in situ without current evidence of active disease, Gleason ≤6 prostate cancer.
* Angina, myocardial infarction symptomatic congestive heart failure, cerebrovascular accident, transient ischemic attack, arterial embolism, pulmonary embolism, percutaneous angioplasty or coronary arterial bypass surgery within the past 3 months.
* History of gastrointestinal perforation or fistula in the past 6 months, or while previously on antiangiogenic therapy, unless underlying risk has been resolved (e.g. through surgical resection or repair).
* The patient has known hypersensitivity to gelatin or lactose monohydrate.
* The patient has received any investigational drug within 28 days prior to registration or 5 half-lives of the investigational drug, whichever is shorter.
* History of bleeding disorders (e.g. pulmonary hemorrhage, significant hemoptysis, menometrorrhagia not responding to hormonal treatment) ≤ 6 weeks before Cycle 1 Day1.
* The patient is on a chronic daily medication known to be a severe or moderate inhibitor or inducer by Micromedex of CYP1A2, CYP2C8, or CYP3A4 at registration.
* Systemic corticosteroids greater than the equivalent of 10 mg of prednisone or equivalent alternative steroid (except physiologic dose for adrenal replacement therapy) or other immunosuppressive agents (such as cyclosporine or methotrexate) and any other medications that could potentially impact the efficacy or safety of the study as judged by the treating investigator are NOT permitted from time of registration to subjects completing protocol therapy unless clinically indicated to manage adverse events or life threatening or serious conditions as determined by the treating investigator.
* Have any condition that, in the opinion of the investigator, would compromise the ability of the subject to meet or perform study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-04-11 (Actual); Primary Completion 2022-10-18 (Actual); Study Completion 2022-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajjai Alva, MD, Principal Investigator — Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ESK981 and Nivolumab: ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Nivolumab: 480 mg/dose IV, Day 1 of each 28-day cycle
  ESK981: ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Nivolumab: 480 mg/dose IV, Day 1 of each 28-day cycle
Period: Overall Study
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab
Started | 8 | 0
Completed | 8 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: No patients were enrolled in the ESK984 and Nivolumab combo arm
Groups:
- Total: Total of all reporting groups
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab | Total
Number analyzed (Participants) | 8 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 4 |  | 4
  >=65 years | 4 |  | 4
Age, Continuous [Median (Full Range); unit: years] | 66 [43 to 78] |  | 66 [43 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 |  | 3
  Male | 5 |  | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0
  Not Hispanic or Latino | 7 |  | 7
  Unknown or Not Reported | 1 |  | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 0 |  | 0
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 7 |  | 7
  More than one race | 0 |  | 0
  Unknown or Not Reported | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 8 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: 1. The Percentage of Patients That Respond to Treatment With the Combination of ESK981 Monotherapy and Nivolumab Therapy (Cohort B).
Description: The percentage of patients in Cohort B that achieve a complete response (CR) or partial response (PR). Response will be assessed by combined Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 and Immune-related (ir)RECIST.
Time Frame: Up to 24 months after last dose of study treatment
Population: No patients were enrolled in the ESK984 and Nivolumab combo arm (cohort B)
Groups:
- ESK981 and Nivolumab (Cohort B): ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Nivolumab: 480 mg/dose IV, Day 1 of each 28-day cycle
  ESK981: ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  Nivolumab: 480 mg/dose IV, Day 1 of each 28-day cycle
Arm/Group | ESK981 and Nivolumab (Cohort B)
Number analyzed (Participants) | 0

2. Secondary Outcome: The Percentage of Patients That Respond to Treatment With ESK981 Monotherapy (Cohort A).
Description: The percentage of patients in Cohort A that achieve a complete response (CR) or partial response (PR). Response will be assessed by RECIST v1.1.
Time Frame: Up to 24 months after last dose of study treatment, 5 month treatment duration on average, no CR or PR responses were recorded.
Measure: Count of Participants; unit: Participants
Groups:
- ESK981 Monotherapy (Cohort A): ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
  ESK981: ESK981: 160 mg (4 capsules) PO daily for 5 consecutive days followed by a 2-day off drug in each week, repeated weekly in 4-week (28-day) cycles
Arm/Group | ESK981 Monotherapy (Cohort A)
Number analyzed (Participants) | 8
Participants | 0

3. Secondary Outcome: Median Overall Survival Time
Description: Overall survival time measured from start of treatment until up to 24 months after the last dose of study treatment in Cohort A (ESK981 monotherapy) and in Cohort B (combination of ESK981 and nivolumab therapy).
Time Frame: Up to 24 months after last dose of study treatment
Population: No patients were enrolled in the ESK984 and Nivolumab combo arm (cohort B)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab
Number analyzed (Participants) | 8 | 0
Months | 24.5 [14.6 to NA] — All the dispersion measures cannot be estimated as we have too few patients. Per PI, there were insufficient number of participants with events to properly measure |

4. Secondary Outcome: Progression Free Survival Time
Description: Measured from start of treatment to time of progression or death, or up to 24 months after the last dose of study treatment in Cohort A (ESK981 monotherapy) and in Cohort B (combination of ESK981 and nivolumab therapy). Disease progression will be assessed by RECIST v1.1 in Cohort A and by combined RECIST v1.1/irRECIST in Cohort B.
Time Frame: Up to 24 months after last dose of study treatment
Population: No patients were enrolled into the combo arm (cohort B)
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab
Number analyzed (Participants) | 8 | 0
months | 1.7 [1.6 to 8.1] |

5. Secondary Outcome: Duration of Therapy
Description: Measured from the first to the last dose of study treatment in Cohort A (ESK981 monotherapy) and in Cohort B (combination of ESK981 and nivolumab therapy).
Time Frame: Up to approximately 24 months after treatment start
Population: No patients were enrolled into the combo arm (cohort B)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab
Number analyzed (Participants) | 8 | 0
Months | 2.1 [0.6 to 19.4] |

6. Secondary Outcome: Duration of Response
Description: Measured from the time of complete response (CR) or partial response (PR) (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Response will be assessed by RECIST v1.1 (Cohort A) and by combined RECIST v1.1/irRECIST (Cohort B).
Time Frame: Up to 24 months after last dose of study treatment
Population: There were no responses to therapy
Arm/Group | ESK981 Monotherapy | ESK981 and Nivolumab
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: All adverse event data (serious and non-serious) collected from the time of the initial study treatment administration through 60 days after the last dose of study drug treatment. Data as collected for 2.5 years
Description: No subjects were enrolled in Cohort B
Arm/Group | ESK981 Monotherapy (Cohort A) | ESK981 and Nivolumab (Cohort B)
All-Cause Mortality (participants affected / at risk) | 3/8 | 0/0
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/0
Other Adverse Events (participants affected / at risk) | 8/8 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESK981 Monotherapy (Cohort A) (N=8) | ESK981 and Nivolumab (Cohort B) (N=0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lung Infection (Infections and infestations) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ESK981 Monotherapy (Cohort A) (N=8) | ESK981 and Nivolumab (Cohort B) (N=0)
Adrenal Insufficiency (Endocrine disorders) | 1 (1) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Alkaline Phosphatase Increased (Investigations) | 2 (2) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 2 (4) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Aspartate Aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 3 (4) | 0 (0)
Bone Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
CD4 Lymphocytes decreased (Investigations) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Creatinine Increase (Investigations) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0)
dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 0 (0)
Flushing (Vascular disorders) | 1 (1) | 0 (0)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
hypertenstion (Vascular disorders) | 2 (3) | NA
joint effusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Localized Edema (General disorders) | 1 (1) | 0 (0)
muscle cramp (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
myalgia (Musculoskeletal and connective tissue disorders) | 2 (3) | 0 (0)
nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Oral Dysesthesia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral Pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (5) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Parethesia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash Maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0)
Thyroid Stimulating Hormone Increased (Investigations) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (3) | 0 (0)
weight loss (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
bilateral ear fullness (Ear and labyrinth disorders) | 1 (1) | 0 (0)
C3-C4 Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
osteopenia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Bladder Mass
peripheral arterial disease (Vascular disorders) | 1 (1) | 0 (0)
right common femoral artery narrowing (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-08-07): https://cdn.clinicaltrials.gov/large-docs/07/NCT03562507/Prot_SAP_000.pdf
  • Informed Consent Form (2019-02-14): https://cdn.clinicaltrials.gov/large-docs/07/NCT03562507/ICF_001.pdf